CLINICAL TRIAL: NCT07095764
Title: Effects of In-Hospital Cardiac Rehabilitation and Manual Lymphatic Drainage in Acute Decompensated Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other); Yeditepe University (Other); Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Melih Zeren, Associate Professor, Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: bakircaymzeren08
Record Dates: First submitted 2025-06-19; First posted 2025-07-31 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-06

CONDITIONS: Acute Decompensated Heart Failure
MeSH Terms: interventions — Manual Lymphatic Drainage; Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Lymphatic Drainage + Cardiac Rehabilitation Group (Experimental): Manual lymphatic drainage and exercise based cardiac rehabilitation will be applied to this group during the hospital stay every day for 3 times a day.
  Interventions: Other: Manual Lymphatic Drainage; Other: Cardiac Rehabilitation
- Cardiac Rehabilitation Group (Active Comparator): Exercise based cardiac rehabilitation will be applied to this group during the hospital stay every day for 3 times a day.
  Interventions: Other: Cardiac Rehabilitation

INTERVENTIONS:
Other: Manual Lymphatic Drainage — Specific manual lymph drainage techniques including stationary circles, rotary circles, pumping, and scooping will be applied to both lower extremities using gentle, rhythmic skin movements in accordance with the direction of the lymphatic flow.
  Arms: Manual Lymphatic Drainage + Cardiac Rehabilitation Group
Other: Cardiac Rehabilitation — An individualized program consists of progressive, low-intensity exercises including respiratory exercises, range of motion exercises for major joints, postural exercises, flexibility exercises, and gradual mobilization exercises such as sitting and walking will be applied.

SUMMARY:
Heart failure is a major global health issue requiring effective interventions to enhance patients' physical function and quality of life. Cardiac rehabilitation, particularly when started early during hospitalization for acute decompensated heart failure, has been shown to improve cardiovascular function, reduce hospital readmissions, and boost recovery. In-hospital exercise training enhances physical capacity, strengthens heart function, and alleviates physical limitations. On the other hand, lymphatic dysfunction in heart failure may also contribute to fluid retention, worsening the symptoms including lower extremity edema. Manual lymphatic drainage is considered a safe method to reduce edema and support fluid balance. This study aims to evaluate effects of in-hospital cardiac rehabilitation and manual lymphatic drainage on fluid overload symptoms and functional capacity in patients with acute decompensated heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized with a diagnosis of acute decompensated heart failure
* Being clinically stable

Exclusion Criteria:

* Having diagnosed pulmonary, neurological, renal, liver, gastrointestinal, orthopedic or oncological pathologies
* Having cardiomyopathy or congestive pericarditis
* Recent heart surgery in the past 6 months
* New or suspected thromboembolic event
* Presence of open wounds, ulcerations or major dermatological diseases in the lower extremities

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-08-12 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Lower extremity edema | At baseline and at hospital discharge, up to 14 days after admission
  Lower extremity edema will be evaluated by circumference measurement
Lower extremity edema | At baseline and at hospital discharge, up to 14 days after admission
  Lower extremity edema will be evaluated by pitting test
Functional capacity | At baseline and at hospital discharge, up to 14 days after admission
  Functional capacity will be measured using 6-min Walk Test.

SECONDARY OUTCOMES:
Health-related quality of life | At baseline and at hospital discharge, up to 14 days after admission
  Health-related quality of life will be evaluted using Short-Form 12 Questionnaire. It is scored between 0-100 and higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University- Cerrahpasa, Cardiology Institute, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided